CLINICAL TRIAL: NCT00986102
Title: A Prospective Study on the Usage Patterns of Doripenem in the Asia Pacific Region
Brief Title: PROUD Study: A Prospective Study on the Usage Patterns of Doripenem in the Asia Pacific Region
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Johnson & Johnson (Hong Kong) Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016321; DORIBAC4007 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2009-09-25; First posted 2009-09-29 (Estimated); Results first posted 2013-02-07 (Estimated); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Pneumonia; Pneumonia, Ventilator-Associated; Urinary Tract Infections
Keywords: Carbapenem; Doripenem; Doribax; Nosocomial pneumonia, Intra-abdominal infections; Urinary tract infection
MeSH Terms: conditions — Pneumonia; Pneumonia, Ventilator-Associated; Urinary Tract Infections; Healthcare-Associated Pneumonia; Intraabdominal Infections | interventions — Doripenem

STUDY DESIGN:
Oversight: FDA-regulated Drug: No

ARMS (1):
- 001 (Other): doripenem 500mg vial by injection every 8 hours for 5 to 14 days
  Interventions: Drug: doripenem

INTERVENTIONS:
Drug: doripenem — 500mg vial by injection every 8 hours for 5 to 14 days

SUMMARY:
The purpose of this study is to understand the utilization patterns of doripenem in Asia Pacific, including the profile of the patients treated with carbapenems.

DETAILED DESCRIPTION:
This is a Phase 4, prospective, open-label, non-comparative, multicenter study to characterize the usage of doripenem in selected hospitals in the Asia Pacific region. Doripenem belongs to the carbapenem class which is a broad-spectrum antibiotic given to treat patients with serious infections, such as pneumonia and complicated intra-abdominal infections. Physicians in the selected hospital or hospital unit will refer potential patients to the study team. Patients will include men and women 18 years of age and older, hospitalized either in the Intensive Care Unit (ICU) or ward, with a diagnosis of pneumonia, complicated intra-abdominal infections and complicated urinary tract infections. The study has 3 phases: a pretreatment phase with a 1-day screening/baseline visit, a treatment phase of 5 to 14 days, and a post-treatment phase consisting of an end-of-treatment (EOT)/early withdrawal visit to be conducted within 24 hours after the last dose of antimicrobial therapy, a test of cure (TOC) visit 7 to 14 days after EOT, a Day 28 visit, and a post-discharge visit 28 days after discharge from the hospital. Usage of Doripenem in terms of approved indications, mode of usage, duration of antibiotic therapy, and patient characteristics will be assessed. Safety will be assessed through monitoring for adverse events, serial physical examinations, and the collection of conventional laboratory data (chemistry panel, complete blood count with differential). Being a prospective study, patient data will be gathered as the patients are enrolled, starting with their present condition and following them until duration of the study. The study will not compare Doripenem with other antibiotics for the primary endpoint. One vial (500mg) of doripenem intravenously (by injection) every 8 hours for 5 to 14 days

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized either in the ICU or ward, with a diagnosis of pneumonia, complicated abdominal infections, or complicated urinary tract infection using the protocol-defined Guidelines for Diagnosis

Exclusion Criteria:

* Pregnant or lactating females
* Allergies to Doripenem or its derivatives
* Infected by a bacteria that is resistant to Doripenem
* Taking probenecid
* Severe allergies to other antibiotics like penicillins, cephalosporins, or carbapenems
* Severe kidney disease, in an unstable disease state and assessed as unlikely to survive until the study follow up period
* Signs of severe sepsis with treatment failure with other carbapenems, who received other carbapenem within 2 weeks before first dose of study drug, and who has any condition that, in the opinion of the investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2009-07-17 (Actual); Primary Completion 2011-09-05 (Actual); Study Completion 2011-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (16):
- Hong Kong, Hong Kong
- Indonesia (3):
  - Bandung
  - Jakarta
  - Surabaya
- Malaysia (9):
  - Ipoh
  - Johor Bahru
  - Kota Bharu
  - Kuala Lumpur
  - Kuala Lumpur K Lumpur
  - Kuala Selangor
  - Pulau Pinang
  - Seremban
  - Terengganu
- Singapore, Singapore
- Vietnam (2):
  - Hanoi
  - Ho Chi Minh City

REFERENCES:
- [Derived] Mustafa M, Chan WM, Lee C, Harijanto E, Loo CM, Van Kinh N, Anh ND, Garcia J. A PROspective study on the Usage patterns of Doripenem in the Asia-Pacific region (PROUD study). Int J Antimicrob Agents. 2014 Apr;43(4):353-60. doi: 10.1016/j.ijantimicag.2014.01.017. Epub 2014 Feb 15. PMID 24636429

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 217 patients were enrolled at sites in Malaysia, Indonesia, Singapore, Vietnam and Hong Kong.
Pre-assignment Details: 217 patients were enrolled and 216 received study medication. 1 patient was enrolled but subsequently withdrew consent before receiving the study medication. 61 patients discontinued study medication prior to end of treatment.
Groups:
- Nosocomial Pneumonia (NP); Ventilator-Associated Pneumonia (VAP): 500 mg of doripenem was administered every 8 hours as 1 or 4-hour infusion for 7 to 14 days
- Complicated Urinary Tract Infection (cUTI): 500 mg of doripenem was administered every 8 hours as 1-hour infusion for 5 to 14 days
- Complicated Intra-abdominal Infection (cIAI): 500 mg of doripenem was administered every 8 hours as 1-hour infusion for 10 days
Period: Overall Study
Arm/Group | Nosocomial Pneumonia (NP) | Ventilator-Associated Pneumonia (VAP) | Complicated Urinary Tract Infection (cUTI) | Complicated Intra-abdominal Infection (cIAI)
Started | 53 (Number of participants who received study medication) | 77 (Number of participants who received study medication) | 19 (Number of participants who received study medication) | 67 (Number of participants who received study medication)
Completed | 52 | 75 | 19 | 66
Not Completed | 1 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nosocomial Pneumonia (NP) | Ventilator-Associated Pneumonia (VAP) | Complicated Urinary Tract Infection (cUTI) | Complicated Intra-abdominal Infection (cIAI) | Total
Number analyzed (Participants) | 53 | 77 | 19 | 67 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (17.52) | 44.4 (19.17) | 58.2 (13.23) | 49.2 (16.13) | 49.5 (17.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 13 | 24 | 72
  Male | 37 | 58 | 6 | 43 | 144
Race/Ethnicity, Customized [Number; unit: Participants]
  Chinese | 8 | 13 | 7 | 28 | 56
  Malay | 33 | 44 | 8 | 35 | 120
  Indian | 2 | 3 | 2 | 0 | 7
  Aboriginal | 0 | 0 | 0 | 1 | 1
  White | 0 | 1 | 0 | 1 | 2
  Others | 10 | 16 | 2 | 2 | 30
Patient's location in the hospital upon enrollment [Number; unit: Participants]
  Intensive Care Unit (ICU) | 30 | 69 | 9 | 29 | 137
  Non -ICU | 23 | 8 | 10 | 36 | 77
  Missing | 0 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Usage of Doripenem as Per the Approved Indication
Description: Early onset of Nosocomial Pneumonia (NP) and Ventilator-Associated Pneumonia (VAP) is defined as less than 5 days after hospitalization and late onset of NP and VAP is defined as more than or equal to 5 days after hospitalization
Time Frame: 5 to 14 days
Population: Intent-to-treat (ITT) population: Included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Nosocomial Pneumonia (NP) | Ventilator-Associated Pneumonia (VAP) | Complicated Urinary Tract Infection (cUTI) | Complicated Intra-abdominal Infection (cIAI)
Number analyzed (Participants) | 53 | 77 | 19 | 67
Participants
  Early onset of NP | 23 | 0 | 0 | 0
  Late onset of NP | 30 | 0 | 0 | 0
  Early onset of VAP | 0 | 32 | 0 | 0
  Late onset of VAP | 0 | 45 | 0 | 0
  Acute Pyelonephritis | 0 | 0 | 11 | 0
  Emphysematous Pyelonephritis | 0 | 0 | 1 | 0
  Prostate Infection | 0 | 0 | 1 | 0
  Pyelonephritis | 0 | 0 | 1 | 0
  Pyonephrosis | 0 | 0 | 1 | 0
  Urosepsis | 0 | 0 | 2 | 0
  Complicated lower urinary tract infection | 0 | 0 | 2 | 0
  Abdominal Abscess | 0 | 0 | 0 | 2
  Appendiceal Abscess | 0 | 0 | 0 | 1
  Appendicitis | 0 | 0 | 0 | 1
  Appendicitis Perforated | 0 | 0 | 0 | 24
  Cholecystitis Acute | 0 | 0 | 0 | 1
  Diverticular Perforation | 0 | 0 | 0 | 2
  Duodenal Ulcer Perforation | 0 | 0 | 0 | 1
  Gallbladder Empyema | 0 | 0 | 0 | 1
  Gastric Perforation | 0 | 0 | 0 | 4
  Gastric Ulcer Perforation | 0 | 0 | 0 | 3
  Gastrointestinal Anastomotic Leak | 0 | 0 | 0 | 2
  Gastrointestinal Stoma Complication | 0 | 0 | 0 | 1
  Ileal Perforation | 0 | 0 | 0 | 2
  Intestinal Perforation | 0 | 0 | 0 | 8
  Large Intestine Perforation | 0 | 0 | 0 | 7
  Pelvic Abscess | 0 | 0 | 0 | 1
  Peritonitis | 0 | 0 | 0 | 1
  Post Procedural Bile Leak | 0 | 0 | 0 | 1
  Small Intestinal Perforation | 0 | 0 | 0 | 3
  Small Intestine Gangrene | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Different Mode of Usage of Doripenem
Time Frame: 5 to 14 days
Population: Intent-to-treat (ITT) population: Included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Nosocomial Pneumonia (NP) | Ventilator-Associated Pneumonia (VAP) | Complicated Urinary Tract Infection (cUTI) | Complicated Intra-abdominal Infection (cIAI)
Number analyzed (Participants) | 53 | 77 | 19 | 67
Participants
  Monotherapy | 41 | 66 | 18 | 62
  Combination Therapy | 12 | 11 | 1 | 5
  First Line Therapy | 16 | 33 | 3 | 30
  Second Line Therapy | 37 | 44 | 16 | 37

3. Primary Outcome: Duration of Antibiotic Therapy
Description: Duration of doripenem and duration of doripenem plus oral antibiotics therapy
Time Frame: 5 to 14 days
Population: Intent-to-treat (ITT) population: Included all enrolled participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Nosocomial Pneumonia (NP) | Ventilator-Associated Pneumonia (VAP) | Complicated Urinary Tract Infection (cUTI) | Complicated Intra-abdominal Infection (cIAI)
Number analyzed (Participants) | 53 | 77 | 19 | 67
Days
  Duration of doripenem therapy | 7.4 (3.51) | 9.2 (4.67) | 6.9 (2.46) | 6.9 (2.86)
  Duration of doripenem plus oral antibiotic therapy | 7.5 (3.57) | 9.9 (6.07) | 9.1 (3.94) | 8.3 (4.50)

4. Primary Outcome: Number of Participants With Acute Physiology and Chronic Health Evaluation II (APACHE II) Score
Description: APACHE II is a severity of disease classification system and the score will be determined in the participants admitted to the Intensive Care Unit upon study enrollment to help predict the risk of mortality for critically ill patients. It consists of, A: acute physiology score (APS; range, 0 to 4), B: age points (range, 0 [less than or equal to 44] to 6 [greater than or equal to 75]) and C: chronic health points (2 [elective postoperative patient] and 5 [non-operative or emergency postoperative patient]). Total APACHE II score is sum of A, B and C.
Time Frame: Baseline (Day -1)
Population: Intent-to-treat (ITT) population: Included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Nosocomial Pneumonia (NP) | Ventilator-Associated Pneumonia (VAP) | Complicated Urinary Tract Infection (cUTI) | Complicated Intra-abdominal Infection (cIAI)
Number analyzed (Participants) | 53 | 77 | 19 | 67
Participants
  APACHE II score: less than or equal to 14 | 34 | 50 | 11 | 58
  APACHE II score: 15 to 19 | 8 | 15 | 3 | 6
  APACHE II score: 20 to 24 | 4 | 7 | 1 | 2
  APACHE II score: 25 to 29 | 2 | 4 | 0 | 0
  APACHE II score: greater than or equal to 30 | 1 | 1 | 0 | 0
  Missing | 4 | 0 | 4 | 1

5. Secondary Outcome: Number of Participants Who Achieved Clinical Cure, Clinical Failure and Intermediate Outcome at End-of-treatment Visit (EOT)
Time Frame: Day 5 or Day 7 or Day 14
Population: Intent-to-treat (ITT) population: Included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Nosocomial Pneumonia (NP) | Ventilator-Associated Pneumonia (VAP) | Complicated Urinary Tract Infection (cUTI) | Complicated Intra-abdominal Infection (cIAI)
Number analyzed (Participants) | 53 | 77 | 19 | 67
Participants
  Clinical cure | 33 | 49 | 15 | 46
  Clinical failure | 7 | 7 | 2 | 6
  Indeterminate outcome | 5 | 15 | 1 | 10
  Missing data | 8 | 6 | 1 | 5

6. Secondary Outcome: Number of Participants Who Achieved Clinical Cure, or Experienced Clinical Failure, Relapse or Intermediate Outcome at Test-of-cure (TOC) Visit
Time Frame: End-of-treatment (Day 5 or Day 7 or Day 14) plus 7 to 14 days
Population: Intent-to-treat (ITT) population: Included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Nosocomial Pneumonia (NP) | Ventilator-Associated Pneumonia (VAP) | Complicated Urinary Tract Infection (cUTI) | Complicated Intra-abdominal Infection (cIAI)
Number analyzed (Participants) | 53 | 77 | 19 | 67
Participants
  Clinical cure | 25 | 39 | 12 | 46
  Clinical failure | 1 | 5 | 2 | 3
  Relapse | 1 | 5 | 1 | 0
  Indeterminate outcome | 4 | 8 | 1 | 4
  Missing data | 22 | 20 | 3 | 14

7. Secondary Outcome: Number of Participants Who Experienced Eradication, Presumed Eradication, Persistence, Presumed Persistence and Indeterminate Response at End-of-treatment Visit (EOT) Visit
Time Frame: Day 5 or Day 7 or Day 14
Population: Microbiological Modified Intent-to-Treat Population (mMITT): included participants who had a baseline pathogen identified, regardless of susceptibility to study medication.
Measure: Number; unit: Participants
Arm/Group | Nosocomial Pneumonia (NP) | Ventilator-Associated Pneumonia (VAP) | Complicated Urinary Tract Infection (cUTI) | Complicated Intra-abdominal Infection (cIAI)
Number analyzed (Participants) | 26 | 63 | 10 | 42
Participants
  Eradication | 7 | 12 | 3 | 7
  Presumed eradication | 10 | 18 | 4 | 18
  Persistence | 0 | 14 | 1 | 0
  Presumed persistence | 3 | 4 | 0 | 3
  Indeterminate | 3 | 10 | 2 | 9
  Missing data | 3 | 5 | 0 | 5

8. Secondary Outcome: Medical Resource Utilization
Description: Medical resource utilization included length of hospital stay, length of intensive care unit (ICU) stay, duration of mechanical ventilation and time to discharge.
Time Frame: From Baseline (Day -1) upto the duration of hospital stay of a participant
Population: Intent-to-treat (ITT) population: Included all enrolled participants who received at least one dose of study medication.
Measure: Median (Full Range); unit: Days
Arm/Group | Nosocomial Pneumonia (NP) | Ventilator-Associated Pneumonia (VAP) | Complicated Urinary Tract Infection (cUTI) | Complicated Intra-abdominal Infection (cIAI)
Number analyzed (Participants) | 53 | 77 | 19 | 67
Days
  Length of hospital stay | 21 (25.89) [3 to 138] | 33 (26.95) [5 to 132] | 13 (12.19) [7 to 53] | 12 (17.60) [5 to 80]
  Length of Intensive Care Unit (ICU) Stay | 8 (14.40) [2 to 54] | 17 (16.34) [3 to 66] | 4 (9.76) [2 to 27] | 7 (10.21) [1 to 52]
  Duration of Mechanical Ventilation | 6 (11.88) [1 to 46] | 15 (21.61) [3 to 115] | 2 (1.92) [1 to 6] | 4 (9.30) [1 to 44]
  Time to Discharge | 13 (15.23) [1 to 63] | 19 (18.96) [1 to 97] | 8 (7.72) [3 to 35] | 9 (16.42) [2 to 88]

9. Secondary Outcome: Number of Participants Readmitted to the Intensive Care Unit (ICU) Within 28 Days After End-of-treatment (EOT)
Time Frame: Within 28 days after EOT (Day 5 or Day 7 or Day 14)
Population: Intent-to-treat (ITT) population: Included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Nosocomial Pneumonia (NP) | Ventilator-Associated Pneumonia (VAP) | Complicated Urinary Tract Infection (cUTI) | Complicated Intra-abdominal Infection (cIAI)
Number analyzed (Participants) | 8 | 19 | 1 | 6
Participants
  Participant still in hospital | 8 | 19 | 1 | 6
  Participant readmitted in ICU | 0 | 1 | 0 | 0

10. Secondary Outcome: Number of Participants Readmitted to the Hospital Within 28 Days After End-of-treatment (EOT)
Time Frame: Within 28 days after EOT (Day 5 or Day 7 or Day 14)
Population: Intent-to-treat (ITT) population: Included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Nosocomial Pneumonia (NP) | Ventilator-Associated Pneumonia (VAP) | Complicated Urinary Tract Infection (cUTI) | Complicated Intra-abdominal Infection (cIAI)
Number analyzed (Participants) | 30 | 44 | 18 | 54
Participants
  Participants discharged from hospital | 30 | 44 | 18 | 54
  Participants readmitted to hospital | 2 | 4 | 1 | 0

ADVERSE EVENTS:
Time Frame: From the time a signed and dated informed consent form is obtained until 30 days after the last dose of study medicaton.
Arm/Group | Nosocomial Pneumonia (NP) | Ventilator-Associated Pneumonia (VAP) | Complicated Urinary Tract Infection (cUTI) | Complicated Intra-abdominal Infection (cIAI)
Serious Adverse Events (participants affected / at risk) | 22/53 | 24/77 | 3/19 | 15/67
Other Adverse Events (participants affected / at risk) | 27/53 | 38/77 | 11/19 | 32/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nosocomial Pneumonia (NP) (N=53) | Ventilator-Associated Pneumonia (VAP) (N=77) | Complicated Urinary Tract Infection (cUTI) (N=19) | Complicated Intra-abdominal Infection (cIAI) (N=67)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardio-Respiratory Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral Valve Stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Right Ventricular Failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric Ulcer Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multi-Organ Failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal Wall Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 4 (5) | 1 (1) | 4 (4)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 5 (5)
Septic Shock (Infections and infestations) | 6 (6) | 4 (4) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wound Infection Fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endotracheal Intubation Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Operative Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural Hypotension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tracheostomy Malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oxygen Saturation Decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-Traumatic Amnestic Disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Dependence On Respirator (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemodynamic Instability (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nosocomial Pneumonia (NP) (N=53) | Ventilator-Associated Pneumonia (VAP) (N=77) | Complicated Urinary Tract Infection (cUTI) (N=19) | Complicated Intra-abdominal Infection (cIAI) (N=67)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 4 (5) | 1 (1) | 3 (3)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left Ventricular Failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myocardial Ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (3)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Parotid Gland Enlargement (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Acinetobacter Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Candiduria (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes Dermatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nosocomial Infection (Infections and infestations) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Peritoneal Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2) | 4 (5) | 2 (2) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Soft Tissue Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal Bacteraemia (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stenotrophomonas Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Alanine Aminotransferase Increased (Investigations) | 4 (4) | 3 (3) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Bilirubin Conjugated Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Alkaline Phosphatase Increased (Investigations) | 5 (5) | 2 (2) | 1 (1) | 0 (0)
Blood Bicarbonate Increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood Bilirubin Unconjugated Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood Cortisol Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Lactate Dehydrogenase Increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Blood Triglycerides Increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Coagulation Time Prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine Renal Clearance Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-Glutamyltransferase Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 5 (5) | 0 (0) | 0 (0) | 1 (1)
Glomerular Filtration Rate Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematocrit Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver Function Test Abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oxygen Saturation Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Red Blood Cell Count Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminases Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White Blood Cell Count Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluid Overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (5) | 2 (2) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5) | 0 (0) | 0 (0)
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 3 (4) | 1 (1) | 4 (6) | 1 (1)
Withdrawal Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days